CLINICAL TRIAL: NCT03627039
Title: Metformin And Cardiovascular Effectiveness vs SGLT2 (MACES)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michael Fralick, Principal investigator, Brigham and Women's Hospital
Other Study IDs: 123
Record Dates: First submitted 2018-07-30; First posted 2018-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; empagliflozin; dapagliflozin; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Truven: NOTE: In the case there are not enough patients/events data will be included from other databases (e.g., Optum, Medicare)
  Interventions: Drug: SGLT2; Drug: Metformin

INTERVENTIONS:
Drug: SGLT2 — All SGLT2 medications approved prior to 2017 will be included (Canagliflozin, empagliflozin, dapagliflozin (all doses, all of the medications are oral)
  Other Names: Canagliflozin, empagliflozin, dapagliflozin (all doses, all of the medications are oral)
Drug: Metformin — Metformin is the main comparator of interest. In a secondary analysis GLP1 will be the comparator
  Other Names: All doses will be included. Metformin is an oral medication.

SUMMARY:
The objective of this study was to compare the effectiveness of sodium glucose co-transporter 2 (SGLT2) inhibitors relative to metformin for reducing subsequent cardiovascular events in patients with type 2 diabetes mellitus.

The investigators will conduct a population-based, new-user, longitudinal-cohort study using a nationwide US commercial insurance claims database. The investigators will compare adults with diabetes mellitus type 2 over the age of 18 who were newly prescribed an SGLT2 inhibitor or metformin between March 29, 2013 (date of US approval of first SGLT2) and January 1st, 2017 (most recent available data). Patients with diabetes mellitus type 2 will be identified using the International Classification of Diseases, Ninth Revision (ICD-9) and ICD-10 codes. Cohort entry date will be the date of the first prescription for an SGLT2 or metformin. New users of SGLT2 or metformin will be defined as those without a prior prescription for either class of medications, or any other medication for diabetes, in the preceding 180 days.

DETAILED DESCRIPTION:
Baseline Covariates: All covariates will be assessed prior to cohort entry. Covariates will reflect diagnoses and procedures recorded during health encounters, including chronic medical conditions (e.g., hypertension, coronary artery disease), diabetes severity (e.g., hemoglobin A1C, end-organ damage), overall healthcare utilization (e.g., recent hospitalization, emergency department visit), prescriber characteristics (e.g., endocrinologist, general practitioner), and medications (e.g., anti-hypertensives, diuretics).

Statistical analysis Propensity score matching will be used to adjust for confounding. The probability of initiating an SGLT2-inhibitor will be calculated through a multivariable logistic regression model containing all of the baseline covariates. Using this propensity score, patients prescribed an SGLT2 were matched 1:1 with patients prescribed metformin using a caliper of up to 0.1 on the probability scale. Covariate balance between the matched cohorts was assessed using standardized differences. Since laboratory data were not available for all patients, these were not included in the propensity score estimation.

After propensity score matching, proportional hazards models will be used to estimate the incidence rate, hazard ratios and 95% confidence intervals for the primary outcome without further adjustments. Schoenfeld residuals will be plotted to assess the proportional hazards assumption. Predefined sensitivity and subgroup analyses included an intention to treat analysis where the censoring criteria of drug discontinuation, switching or augmentation are removed. The investigators will also assess the primary risk in a cohort restricted to patients with a past-history of cardiovascular disease if our sample size allows it. To test the specificity of our findings, the investigators will also conduct a tracer analysis using cellulitis as an outcome, since cellulitis is not associated with SGLT2s or metformin.

ELIGIBILITY:
INCLUSION:

- all patients newly prescribed an SGLT2 or metformin between March 29, 2013 to January 1st, 2017 with at least 6 months of continuous enrollment (1 year in a sensitivity analysis)

EXCLUSION:

* age < 18 years
* previous use of any diabetes medication
* lack of a diagnosis of type 2 diabetes mellitus
* history of malignant neoplasm
* dialysis
* type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will conduct a population-based, new-user, longitudinal-cohort study using the nationwide US commercial insurance claims database. This database provides patient demographics and longitudinal, individual-level data on healthcare utilization, inpatient and outpatient diagnoses, diagnostic tests, clinical procedures, outpatient laboratory results, and pharmacy dispensing of drugs.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular composite (stroke, myocardial infarction, heart failure) | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  The outcome will be identified using ICD9 and ICD10 codes and reported as rates of acute myocardial infarction, heart failure, stroke (they will only be analyzed individually if there are sufficient number of one of the events defined as > 30 events)

SECONDARY OUTCOMES:
Harms: Hypoglycemia | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  Hypoglycemia: identified using ICD9 and ICD10 codes and reported as rates
Harms: diabetic ketoacidosis | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  Diabetic ketoacidosis: identified using ICD9 and ICD10 codes and reported as rates
Harms: lactic acidosis | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  Lactic acidosis: identified using ICD9 and ICD10 codes and reported as rates
Harms: Acute kidney injury | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  Acute kidney injury: identified using ICD9 and ICD10 codes and reported as rates
Harms: Genital infection | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  Genital infection: identified using ICD9 and ICD10 codes and reported as rates
Costs | Follow-up will begin one day after cohort entry and cost analysis will end 1 year thereafter
  Costs of metformin compared to SGLT2. Estimates for costs associated with the individual outcomes.

OTHER OUTCOMES:
Tracer outcomes | Follow-up will begin one day after cohort entry and continue until medication discontinuation, study outcome, or no further data. Most patients will have 200 days of follow up
  The outcome will be identified using ICD9 and ICD10 codes and reported as rates (1) Cellulitis

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pharmacoepidemiology and Pharmacoeconomics, Boston, Massachusetts, United States